CLINICAL TRIAL: NCT04824885
Title: Study of a Dialysate Without Acetate on Protein Energy Wasting Syndrome in Chronic Hemodialysis Patient
Brief Title: Study of a Dialysate Without Acetate on Protein Energy Wasting Syndrome in Chronic Hemodialysis Patient (EASY)
Acronym: EASY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: INRAE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AOI 2019 ANIORT; 2020-A00678-31 (Other: ANSM)
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease; Hemodialysis
Keywords: Acetate free dialysate; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Equipment and Supplies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetate free then acetate containing dialysate (Experimental): Patients in group 1 will first be treated with the acetate-free dialysate (A-D) for 6 months and then the acetate-containing dialysate (A + D) for 6 months.
  Interventions: Device: Chlorhydric acid based acid concentrate for bicarbonate hemodialysis (medical device)
- Acetate containing dialysate then acetate free dialysate (Experimental): Group 2 patients will continue on the usual dialysate (A + D) for 6 months and then switch to A-D dialysate for the next 6 months. Patients will be blinded from study treatment.
  Interventions: Device: Chlorhydric acid based acid concentrate for bicarbonate hemodialysis (medical device)

INTERVENTIONS:
Device: Chlorhydric acid based acid concentrate for bicarbonate hemodialysis (medical device) — usual dialysate (A + D) for 6 months and then switch to A-D dialysate for the next 6 months

SUMMARY:
This work aims to study the effect of an acetate-free dialysate on protein-energy wasting syndrome in patients with chronic hemodialysis renal failure, in comparison to a conventional dialysate with acetate. The hypothesis is that a dialysate without acetate would improve patients nutritional status

DETAILED DESCRIPTION:
The dialysate usually used at the Clermont Ferrand CHU dialysis center is a dialysate containing acetate After inclusion, patients will be randomly divided into two groups. Patients in group 1 will first be treated with the acetate-free dialysate (A-D) for 6 months and then the acetate-containing dialysate (A + D) for 6 months. Group 2 patients will continue on the usual dialysate (A + D) for 6 months and then switch to A-D dialysate for the next 6 months. Patients will be blinded from study treatment.

Patients will be followed for 1 year.

A the beginning then every 3 months will be carried out:

* A measurement of body composition by multi-frequency bioimpedancemetry
* A measurement of the gripping force by a dynamometer (hand grip force )
* A 4-meter walk test
* A SARC-F Sarcopenia Assessment Questionnaire A blood test for the usual biological analyzes carried out as part of the recommendations for monitoring patients on hemodialysis will be carried out every month.

An additional blood sample (5.5 mL) for quantification of the levels of expression of potential blood biomarkers of muscle condition will be taken initially, at 6 months and at 12 months (i.e. 16.5 mL more compared to current practice). ).

ELIGIBILITY:
Inclusion Criteria:

* Major patient;
* Man or woman ;
* Treated with intermittent hemodialysis for chronic renal failure;
* Affiliated with a social security scheme;
* Having given a signed agreement after detailed explanation of the protocol on the basis of the information sheet and likely to comply with it

Exclusion Criteria:

* Patient with lower limb amputation more proximal than a transmetatarsal amputation (invalidity of the model for estimating body composition by BCM in this situation)
* Acute event in the 3 months preceding inclusion (infection, surgery).
* Having a neuromuscular pathology responsible for a motor deficit.
* Whose life expectancy does not exceed 6 months
* With a psychiatric pathology or cognitive impairment rendering him unable to give informed consent
* Pregnant women
* Patient under guardianship, curatorship or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
prealbumin | change at 6 months from the start of Acetate free or acetate containing dialysate
  biochemical measurement

SECONDARY OUTCOMES:
Muscle mass | change at 6 months from the start of acetate free or acetate containing dialysate
  Lean Tissue Index or LTI from the spectral analysis of body bioimpedance according to the model of Chamney et al, creatine index according Desmeules et al
Muscle performance | change at 6 months from the start of acetate free or acetate containing dialysate
  meter walk test
Muscle performance with hand grip test | change at 6 months from the start of acetate free or acetate containing dialysate
  hand grip test
SARC-F | change at 6 months from the start of acetate free or acetate containing dialysate
  Result of SARC-F survey
muscle biomarkers | Month 6
  blood RNA
muscle biomarkers | Year 1
  blood RNA
mortality | Year 1
  Time to death
morbidity | Year 1
  Time to cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Julien Aniort, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France